



An Evaluation of an ACT and PBS Group for Parents and Education Staff of Children and Young People with an Intellectual Disability
Parent Consent Form (non-CTIMP/CE device), version no. 2, 17/12/2018

## **Consent Form (version 2)**

## An Evaluation of an ACT and PBS Group for Parents and Education Staff of Children and Young People with an Intellectual Disability

| Participant ID: | | | |
|---|---|---|---|
| | | Initial here for YES | Initial here for NO |
| 1. I confirm that I have read and unde | rstand the information sheet (P | arent | |
| PIS version 2, 17.12.2018) for the abo | ve study and have had the | | |
| opportunity to consider the information | for a minimum of 24 hours and | d ask | |
| questions. | | | |
| 2. I understand that my participation is | voluntary and that I am free to | | |
| withdraw at any time, without giving ar | y reason, without my medical o | care or | |
| legal rights being affected. | | | |
| 3. I understand that relevant sections of | of data collected during the stud | dy may | |
| be looked at by individuals from the re- | gulatory authorities and from th | e | |
| Sponsors (NHS Lothian and the Unive | rsity of Edinburgh) or from the/ | other | |
| NHS Board(s) where it is relevant to m | y taking part in this research. I | give | |
| permission for those individuals to hav | e access to my records. | | |
| 4. I agree to my General Practitioner ( | GP) being informed of my partic | cipation | |
| in this study. | | | |
| 5. I agree to a summary of the study re | esults being sent to me by post. | | |
| 6. I agree to the focus group being | audio-recorded, for the purpo | oses of | |
| allowing it to be transcribed. | | | |
| 7. I agree to take part in the above students | dy. | | |
| | | · | |
| Name of Participant | Date | Signature | |
| Name of Person taking consent | <br>Date | Signature | |
| | <del>=</del> | - 3 | |

1x original – into Site File; 1x copy – to Participant;